CLINICAL TRIAL: NCT00404352
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial of Rebif New Formulation (44 Microgram [Mcg] Three Times Weekly [Tiw] and 44 Mcg Once Weekly [ow]) in Subjects at High Risk of Converting to Multiple Sclerosis (REFLEX)
Brief Title: REbif FLEXible Dosing in Early Multiple Sclerosis (MS)
Acronym: REFLEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMP27025; 2006-002982-38 (EudraCT Number)
Record Dates: First submitted 2006-11-27; First posted 2006-11-28 (Estimated); Results first posted 2012-09-24 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-12

CONDITIONS: Multiple Sclerosis
Keywords: Rebif New Formulation; Clinical Isolated Syndrome; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RNF 44 mcg three times weekly (Active Comparator)
  Interventions: Drug: RNF
- RNF 44 mcg once weekly and placebo twice weekly for blinding (Active Comparator)
  Interventions: Drug: RNF; Drug: Placebo
- Placebo three times weekly (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RNF — Single dose of RNF administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months, or 36 months for patients enrolled in the OL extension.
  Other Names: Rebif
  Arms: RNF 44 mcg once weekly and placebo twice weekly for blinding; RNF 44 mcg three times weekly
Drug: RNF — Single dose of RNF administered subcutaneously once weekly at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months.
  Other Names: Rebif
  Arms: RNF 44 mcg once weekly and placebo twice weekly for blinding; RNF 44 mcg three times weekly
Drug: Placebo — Placebo was supplied as a transparent, sterile solution for injection in pre-filled syringes matching the RNF pre-filled syringes, each containing 0.5 mL.
  Arms: Placebo three times weekly; RNF 44 mcg once weekly and placebo twice weekly for blinding

SUMMARY:
The study is a 24 months randomized, double-blind, Placebo-controlled, multi-center clinical trial with an optional 12 months open label extension.

The primary objective of the study is to evaluate the effect of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of Interferon [IFN] beta-1a (RNF) 44 microgram (three times weekly and once weekly) versus placebo on the time to conversion to McDonald multiple sclerosis (MS) criteria (2005) in subjects with a first clinical demyelinating event at high risk of converting to MS.

The main secondary objective of study is to evaluate the effect of RNF 44 microgram (three times weekly and once weekly) versus placebo on the "Time to conversion to clinically definite MS (CDMS)" in subjects with a first clinical demyelinating event at high risk of converting to MS.

At the end of 24 month double-blind core REFLEX trial, subjects who will not convert to CDMS and decide to receive open-label (OL) treatment will be enrolled into an open-label, 12 month extension period to evaluate the effect of RNF 44 mcg three times weekly treatment on the time to conversion to McDonald MS and time to conversion to CDMS.

ELIGIBILITY:
Inclusion Criteria:

* Single, first clinical event suggestive of MS within 60 days prior to study Day 1, which is the day of randomization (clock starts 24 hours after onset). The event must be a new neurological abnormality present for at least 24 hours, either mono- or polysymptomatic, other than a paresthesia, vegetative or cerebral dysfunction
* At least two clinically silent lesions on the T2-weighted MRI scan, with a size of at least 3 millimeter (mm), at least one of which is ovoid or periventricular or infratentorial
* EDSS 0 - 5.0 at least one time point during the screening period before start of treatment
* 18 and 50 years old, inclusive
* Willing to follow study procedures
* Written informed consent
* If female, subject must:

  * be neither pregnant nor breast-feeding nor attempting to conceive
  * use a highly effective method of contraception. A highly effective method of contraception is defined as those which result in a low failure rate (that is [i.e.] less than 1 percent [%] per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomised partner

Exclusion Criteria:

* Diagnosis of MS (per McDonald criteria 2005)
* Any other disease that could better explain the subject's signs and symptoms
* Complete transverse myelitis or bilateral optic neuritis
* Subject uses or has used any other approved MS disease-modifying drug (DMD)
* Any investigational drug or undergone an experimental procedure within 12 weeks prior to study Day 1
* Oral or systemic corticosteroids or adrenocorticotropic hormone (ACTH) within 30 days prior to study Day 1
* Total bilirubin greater than 2.5 times upper limit of normal (ULN)
* Subject has total aspartate aminotransferase (AST) or alanine aminotransferase (ALT) or alkaline phosphatase (ALP) greater than 2.5 times the ULN
* Inadequate bone marrow reserve, defined as a total white blood cell count less than 3.0 x 109 per liter (/L), platelet count less than 75 x 109/L, hemoglobin less than 100 gram per liter (g/L)
* Current autoimmune disease
* Major medical or psychiatric illness (including history of or current severe depressive disorders and/or suicidal ideation) that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
* History of seizures not adequately controlled by treatment
* Cardiac disease, such as angina, congestive heart failure or arrhythmia
* Known allergy to IFN-beta or the excipient(s) of the study medication
* Any condition that could interfere with the MRI evaluation;
* Known allergy to gadolinium-diethylene triamine pentaacetic acid (DTPA)
* Previously participated in this study
* Participated in any clinical trial within the past 6 months
* Any immunomodulatory or immunosuppressive therapy at any time prior to enrollment, including, but not limited to, the following products: any IFN, glatiramer acetate (Copolymer I), cyclophosphamide, cyclosporine, methotrexate, linomide, azathioprine, mitoxantrone, teriflunomide, laquinimod, cladribine, total lymphoid irradiation, anti-lymphocyte monoclonal antibody treatment (e.g. natalizumab, alemtuzumab/Campath, anti-cluster of differentiation 4 [CD4]), intravenous, immunoglobulins (Igs), cytokines or anti-cytokine therapy
* Any experimental MS treatment prior to trial entry, including, but not limited to, any statins (if given to prevent MS) and pentoxyfylline
* History of alcohol or drug abuse
* Intolerance or any contraindication to both paracetamol (acetaminophen) and ibuprofen
* Inability to administer subcutaneous injections either by self or by caregiver
* Moderate to severe renal impairment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 517 (Actual)
Dates: Start 2006-11; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina M. Stubinski, MD, Study Director — Merck Serono S.A., Geneva
Locations (67):
- Research Site, Mendoza, Argentina
- Research Site, Sydney, Australia
- Austria (2):
  - Research Site, Graz
  - Research Site, Innsbruck
- Belgium (2):
  - Research Site, B-Leuven
  - Research Site, Bruges
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Shumen
  - Research Site, Sofia
  - Research Site, Varna
- Canada (3):
  - Research Site, Montreal, Quebec
  - Research Site, Ontario
  - Research Site, Victoria British Columbia
- Croatia (5):
  - Research Site, Karlovac
  - Research Site, Osijek
  - Research Site, Rijeka
  - Research Site, Split
  - Research Site, Zagreb
- Czechia (3):
  - Research Site, Hradec Králové
  - Research Site, Olomouc
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (2):
  - Research Site, OYS
  - Research Site, Vantaa
- France (2):
  - Research Site, Paris
  - Research Site, Poissy
- Germany (3):
  - Research Site, Hanover
  - Research Site, Henningsdorf
  - Research Site, Munich
- Research Site, Athens, Greece
- Israel (3):
  - Research Site, Ness Ziona
  - Research Site, Safed
  - Research Site, Tel Litwinsky
- Italy (4):
  - Research Site, Catania
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Roma
- Research Site, Riga, Latvia
- Research Site, Beirut, Lebanon
- Research Site, Rabat, Morocco
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Lisbon, Portugal
- Romania (4):
  - Research Site, Bucharest
  - Research Site, Iași
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Russia (7):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Saratov
  - Research Site, Yekaterinburg
- Research Site, Riyadh, Saudi Arabia
- Serbia (2):
  - Research Site, Belgrade
  - Research Site, Niš
- Research Site, Prešov, Slovakia
- Spain (4):
  - Research Site, Barcelona
  - Research Site, Bilbao
  - Research Site, Madrid
  - Research Site, Seville
- Research Site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Kuhle J, Leppert D, Comi G, de Stefano N, Kappos L, Freedman MS, Seitzinger A, Roy S. Serum neurofilament light chain correlations in patients with a first clinical demyelinating event in the REFLEX study: a post hoc analysis. Ther Adv Neurol Disord. 2024 Mar 29;17:17562864241239101. doi: 10.1177/17562864241239101. eCollection 2024. PMID 38560407
- [Derived] Battaglini M, Vrenken H, Tappa Brocci R, Gentile G, Luchetti L, Versteeg A, Freedman MS, Uitdehaag BMJ, Kappos L, Comi G, Seitzinger A, Jack D, Sormani MP, Barkhof F, De Stefano N. Evolution from a first clinical demyelinating event to multiple sclerosis in the REFLEX trial: Regional susceptibility in the conversion to multiple sclerosis at disease onset and its amenability to subcutaneous interferon beta-1a. Eur J Neurol. 2022 Jul;29(7):2024-2035. doi: 10.1111/ene.15314. Epub 2022 Apr 4. PMID 35274413
- [Derived] Freedman MS, De Stefano N, Barkhof F, Polman CH, Comi G, Uitdehaag BM, Casset-Semanaz F, Hennessy B, Lehr L, Stubinski B, Jack DL, Kappos L. Patient subgroup analyses of the treatment effect of subcutaneous interferon beta-1a on development of multiple sclerosis in the randomized controlled REFLEX study. J Neurol. 2014 Mar;261(3):490-9. doi: 10.1007/s00415-013-7222-6. Epub 2014 Jan 12. PMID 24413638
- [Derived] De Stefano N, Comi G, Kappos L, Freedman MS, Polman CH, Uitdehaag BM, Hennessy B, Casset-Semanaz F, Lehr L, Stubinski B, Jack DL, Barkhof F. Efficacy of subcutaneous interferon beta-1a on MRI outcomes in a randomised controlled trial of patients with clinically isolated syndromes. J Neurol Neurosurg Psychiatry. 2014 Jun;85(6):647-53. doi: 10.1136/jnnp-2013-306289. Epub 2013 Nov 29. PMID 24292999
- [Derived] Comi G, De Stefano N, Freedman MS, Barkhof F, Polman CH, Uitdehaag BM, Casset-Semanaz F, Hennessy B, Moraga MS, Rocak S, Stubinski B, Kappos L. Comparison of two dosing frequencies of subcutaneous interferon beta-1a in patients with a first clinical demyelinating event suggestive of multiple sclerosis (REFLEX): a phase 3 randomised controlled trial. Lancet Neurol. 2012 Jan;11(1):33-41. doi: 10.1016/S1474-4422(11)70262-9. Epub 2011 Dec 4. Erratum In: Lancet Neurol. 2012 Feb;11(2):125. PMID 22146409
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were recruited in 78 centers across 28 countries for REFLEX study. REFLEX 12 months open label extension (OLE) was conducted at 11 active centers in 9 countries.
Groups:
- RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population): Single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of interferon [IFN]-beta-1a (RNF) injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months or until conversion to clinically definite multiple sclerosis (CDMS) whichever occurs first.
- RNF 44 Mcg Once Weekly (DB Population): Single dose of RNF injection administered subcutaneously once weekly plus 2 matching placebo doses at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months or until conversion to CDMS whichever occurs first.
- Placebo (DB Population): Single dose of matching placebo administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months or until conversion to CDMS whichever occurs first.
- RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly: After having converted to CDMS, participants received open-label (OL) study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months.
- RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly; Placebo/OL RNF 44 Mcg Three Times Weekly: After having converted to CDMS, participants received OL study treatment with RNF. Single dose of RNF injection administrated subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months.
- RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE): Participants who were not converted to CDMS and completed 24 month core REFLEX trial were enrolled in a 1 year open label extension (OLE). Participants who had received RNF three times a week in the core REFLEX trial, were re-titrated with a single dose of RNF injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months in this 12 months open label extension.
- RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE): Participants who were not converted to CDMS and completed 24 month core REFLEX trial were enrolled in a 1 year OLE. Participants who had received RNF once weekly in the core REFLEX trial were re-titrated with a single dose of RNF injection subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months in this 12 months open label extension.
- Placebo/RNF 44 Mcg Three Times Weekly (OLE): Participants who were not converted to CDMS and completed 24 month core REFLEX trial were enrolled in a 1 year OLE. Participants who had received placebo in the core REFLEX trial were re-titrated with a single dose of RNF injection subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 mcg for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 36 months in this 12 months open label extension.
Period: Double Blind (up to 24 Month)
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population) | RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly | RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly | Placebo/OL RNF 44 Mcg Three Times Weekly | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Started | 171 | 175 | 171 | 0 | 0 | 0 | 0 | 0 | 0
Treated | 171 | 173 | 171 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 119 | 128 | 92 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 52 | 47 | 79 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 5 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 8 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Disease progression | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Poor compliance | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Switched to open label phase | 31 | 30 | 59 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Randomized but not treated | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label (up to 24 Month)
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population) | RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly | RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly | Placebo/OL RNF 44 Mcg Three Times Weekly | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Started | 0 | 0 | 0 | 31 (From DB period, 31 participants converted to CDMS and switched to OL period in this study) | 30 (From DB period, 30 participants converted to CDMS and switched to OL period in this study) | 59 (From DB period, 59 participants converted to CDMS and switched to OL period in this study) | 0 | 0 | 0
Completed | 0 | 0 | 0 | 28 | 28 | 52 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 3 | 2 | 7 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Disease progression | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Open Label Extension (up to 36 Months)
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population) | RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly | RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly | Placebo/OL RNF 44 Mcg Three Times Weekly | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 4 (4 participants who did not convert to CDMS in 24 months and gave consent to enroll in OLE period) | 5 (5 participants who did not convert to CDMS in 24 months and gave consent to enroll in OLE period) | 11 (11 participants who did not convert to CDMS in 24 months and gave consent to enroll in OLE period)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population) | Total
Number analyzed (Participants) | 171 | 175 | 171 | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (8.5) | 30.7 (8.1) | 30.9 (7.9) | 30.7 (8.2)
Age, Customized [Number; unit: participants]
  Less than 30 years | 86 | 86 | 87 | 259
  Greater than or equal to 30 years | 85 | 89 | 84 | 258
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 114 | 106 | 112 | 332
  Male | 57 | 69 | 59 | 185
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 0 | 0 | 0
  Black | 0 | 1 | 0 | 1
  White | 171 | 174 | 171 | 516
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Conversion to Multiple Sclerosis (MS) According to the McDonald Criteria (2005)
Description: The McDonald criteria use dissemination in time and space established by magnetic resonance image (MRI) findings to provide a clinical diagnosis for MS. Dissemination in time is established by a new time constant 2 (T2) or gadolinium-enhancing (Gd+) lesion found on a repeat MRI. Dissemination in space is established by the presence of any 3 of the following: 1 Gd+ lesion or 9 T2 bright lesions if there is no enhancement; greater than or equal to 1 infratentorial lesion; greater than or equal to 1 juxtacortical lesion; greater than or equal to 3 periventricular lesions.
Time Frame: Various time points from randomization up to 24 months
Population: Intent-to-treat (ITT) population included all participants who were randomized to the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population)
Number analyzed (Participants) | 171 | 175 | 171
days | 310 [183 to 488] | 182 [107 to 270] | 97 [93 to 101]
Statistical Analysis 1: Comparison: RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) vs Placebo (DB Population); Test type: Superiority or Other; p < 0.001, Log Rank; Log-rank test was stratified for controlling randomization stratification factors
Statistical Analysis 2: Comparison: RNF 44 Mcg Once Weekly (DB Population) vs Placebo (DB Population); Test type: Superiority or Other; p = 0.008, Log Rank; Log-rank test was stratified for controlling randomization stratification factors
Statistical Analysis 3: Comparison: RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) vs RNF 44 Mcg Once Weekly (DB Population); Test type: Superiority or Other; p = 0.009, Log Rank; Log-rank test was stratified for controlling randomization stratification factors

2. Secondary Outcome: Time to Conversion to Clinically Definite Multiple Sclerosis (CDMS) Defined by Either a Second Attack or a 3-Month Sustained Increase (Greater Than or Equal to 1.5 Points) in the Expanded Disability Status Scale (EDSS) Score
Description: CDMS was defined by the occurrence of a second exacerbation or relapse over 24 months in participants who presented with first clinical demyelinating event (FCDE) accompanied by an abnormal MRI scan. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
Time Frame: Various time points from randomization up to 24 months
Population: ITT population included all participants who were randomized to the assigned study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population)
Number analyzed (Participants) | 171 | 175 | 171
days | NA [NA to NA] — Non-estimable: Insufficient participants reached the median percentile to calculate the upper and lower limits of confidence interval. | NA [NA to NA] — Non-estimable: Insufficient participants reached the median percentile to calculate the upper and lower limits of confidence interval. | NA [NA to NA] — Non-estimable: Insufficient participants reached the median percentile to calculate the upper and lower limits of confidence interval.
Statistical Analysis 1: Comparison: RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) vs Placebo (DB Population); Test type: Superiority or Other; p < 0.001, Log Rank; Log-rank test was stratified for controlling randomization stratification factors
Statistical Analysis 2: Comparison: RNF 44 Mcg Once Weekly (DB Population) vs Placebo (DB Population); Test type: Superiority or Other; p = 0.002, Log Rank; Log-rank test was stratified for controlling randomization stratification factors
Statistical Analysis 3: Comparison: RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) vs RNF 44 Mcg Once Weekly (DB Population); Test type: Superiority or Other; p = 0.774, Log Rank; Log-rank test was stratified for controlling randomization stratification factors

3. Secondary Outcome: Time to Conversion to Clinically Definite Multiple Sclerosis (CDMS) Defined by Either a Second Attack or a 3-Month Sustained Increase (Greater Than or Equal to 1.5 Points) in the Expanded Disability Status Scale (EDSS) Score
Description: CDMS was defined by the occurrence of a second exacerbation or relapse over 36 months in participants who presented with FCDE accompanied by an abnormal MRI scan. EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated.
Time Frame: Various time points from randomization up to 36 months
Population: OL ITT population included all participants who were randomized at baseline in core REFLEX trial and entered the 12 months OLE period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Number analyzed (Participants) | 4 | 5 | 11
days | NA [NA to NA] — Insufficient participants reached the median percentile to calculate the upper and lower limits of confidence interval. | NA [NA to NA] — Insufficient participants reached the median percentile to calculate the upper and lower limits of confidence interval. | NA [NA to NA] — Insufficient participants reached the median percentile to calculate the upper and lower limits of confidence interval.

4. Secondary Outcome: Mean Number of Combined Unique Active (CUA) Lesions, New Time Constant 2 (T2) Lesions, Gadolinium Enhanced (Gd+) Lesions and New Time Constant 1 (T1) Hypointense Lesions Per Participant Per Scan
Description: Number of CUA lesions, new T2 lesions, Gd+ lesions and new T1 hypointense lesions were measured by using MRI scans.
Time Frame: Month 24 up to Month 36
Population: OL ITT population included all participants who were randomized at baseline in core REFLEX trial and entered the 12 months OLE period. "n" signifies those participants who were evaluated for this measure at the specified time point for each arm group respectively.
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Number analyzed (Participants) | 4 | 5 | 11
lesions
  CUA lesions (n=3,5,9) | 0.33 (0.58) | 0.00 (0.00) | 1.56 (2.93)
  New T2 lesions (n=3,5,9) | 0.17 (0.29) | 0.00 (0.00) | 0.94 (1.61)
  New Gd+ lesions (n=3,5,9) | 0.17 (0.29) | 0.00 (0.00) | 0.56 (1.21)
  New T1 Hypointense lesions (n=3,5,9) | 0.17 (0.29) | 0.00 (0.00) | 0.56 (0.88)

5. Secondary Outcome: Change From Baseline in Time Constant 2 (T2) Lesion Volume , Time Constant 1 (T1) Hypointense Lesion Volume and Gadolinium Enhanced (Gd+) Lesion Volume at Month 36
Description: Change from baseline in lesion volume was measured by using MRI scans for T2 lesions, T1 hypointense lesions and (Gd+) lesions.
Time Frame: Baseline, Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cubic millimeter (mm^3)
Arm/Group | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Number analyzed (Participants) | 4 | 5 | 11
cubic millimeter (mm^3)
  T2 lesion volume at Baseline (n=4,5,11) | 675.20 (940.87) | 1703.48 (1324.41) | 3533.37 (3914.98)
  T2 lesion volume change at Month 36 (n=2,4,8) | 180.25 (198.34) | -22.63 (382.14) | -1155.63 (3348.36)
  T1 lesion volume at Baseline (n=4,5,11) | 30.05 (60.10) | 302.70 (358.58) | 488.72 (589.06)
  T1 lesion volume change at Month 36 (n=2,4,8) | 55.75 (78.84) | 216.68 (310.06) | 138.89 (339.99)
  Gd+ lesion volume at Baseline (n=4,5,11) | 103.70 (151.17) | 0.00 (0.00) | 287.15 (649.68)
  Gd+ lesion volume change at Month 36 (n=2,4,8) | -47.20 (66.75) | 0.00 (0.00) | -246.08 (848.99)

6. Primary Outcome: Time to Conversion to Multiple Sclerosis (MS) According to the McDonald Criteria (2005)
Description: The McDonald criteria use dissemination in time and space established by MRI findings to provide a clinical diagnosis for MS. Dissemination in time is established by a T2 or Gd+ lesion found on a repeat MRI. Dissemination in space is established by the presence of any 3 of the following: 1 Gd+ lesion or 9 T2 bright lesions if there is no enhancement; greater than or equal to 1 infratentorial lesion; greater than or equal to 1 juxtacortical lesion; greater than or equal to 3 periventricular lesions.
Time Frame: Various time points from randomization up to 36 months
Population: Open label (OL) ITT population included all participants who were randomized at baseline in core REFLEX trial and entered the 12 months OLE period.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Number analyzed (Participants) | 4 | 5 | 11
days | NA [NA to NA] — Data could not be analyzed as none of the participants converted to MS according to the McDonald Criteria in the 12 month OLE period. | NA [NA to NA] — Data could not be analyzed as none of the participants converted to MS according to the McDonald Criteria in the 12 month OLE period. | NA [NA to NA] — Data could not be analyzed as none of the participants converted to MS according to the McDonald Criteria in the 12 month OLE period.

7. Secondary Outcome: Change From Baseline in Expanded Disability Status Score (EDSS) Score at Month 36
Description: EDSS assesses disability in 8 functional systems. An overall score ranging from 0 (normal) to 10 (death due to MS) was calculated. The change in EDSS at Month 36 was calculated as EDSS at Month 36 minus EDSS at baseline.
Time Frame: Baseline, Month 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Number analyzed (Participants) | 4 | 5 | 11
unit on a scale
  Baseline (n=4,5,11) | 1.88 (0.85) | 1.60 (0.96) | 1.64 (0.67)
  Change at Month 36 (n=2,4,8) | -0.25 (1.06) | -0.63 (0.48) | -0.50 (0.65)

ADVERSE EVENTS:
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Groups:
- RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population): Single dose of fetal bovine serum [FBS]-free/human serum albumin [HSA]-free formulation of interferon [IFN]-beta-1a (RNF) injection administered subcutaneously three times weekly at least 48 hours apart at a starting dose of 8.8 microgram (mcg) for first 2 weeks followed by 22 mcg for next 2 weeks and finally 44 mcg until 24 months or until conversion to CDMS whichever occurs first.
Arm/Group | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) | RNF 44 Mcg Once Weekly (DB Population) | Placebo (DB Population) | RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly | RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly | Placebo/OL RNF 44 Mcg Three Times Weekly | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) | Placebo/RNF 44 Mcg Three Times Weekly (OLE)
Serious Adverse Events (participants affected / at risk) | 6/171 | 8/173 | 12/171 | 1/31 | 0/30 | 1/59 | 0/4 | 0/5 | 0/11
Other Adverse Events (participants affected / at risk) | 149/171 | 156/173 | 133/171 | 20/31 | 20/30 | 47/59 | 3/4 | 2/5 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) (N=171) | RNF 44 Mcg Once Weekly (DB Population) (N=173) | Placebo (DB Population) (N=171) | RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly (N=31) | RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly (N=30) | Placebo/OL RNF 44 Mcg Three Times Weekly (N=59) | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) (N=4) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) (N=5) | Placebo/RNF 44 Mcg Three Times Weekly (OLE) (N=11)
Appendicitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Varicella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Post procedural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Deafness congenital (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Dermoid cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Iron deficiency anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Ischemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RNF 44 Mcg Three Times Weekly (Double Blind [DB] Population) (N=171) | RNF 44 Mcg Once Weekly (DB Population) (N=173) | Placebo (DB Population) (N=171) | RNF 44 Mcg Three Times Weekly/OL RNF 44 Mcg Three Times Weekly (N=31) | RNF 44 Mcg Once Weekly/OL RNF 44 Mcg Three Times Weekly (N=30) | Placebo/OL RNF 44 Mcg Three Times Weekly (N=59) | RNF 44Mcg Three Times Weekly/RNF 44Mcg Three Times Weekly(OLE) (N=4) | RNF 44 Mcg Once Weekly/RNF 44 Mcg Three Times Weekly (OLE) (N=5) | Placebo/RNF 44 Mcg Three Times Weekly (OLE) (N=11)
Influenza like illness (General disorders) | 93 (218) | 122 (374) | 34 (50) | 8 (9) | 3 (6) | 24 (31) | 1 | 1 | 1
Injection site erythema (General disorders) | 50 (76) | 34 (49) | 3 (3) | 4 (5) | 3 (5) | 13 (13) | 0 | 0 | 0
Pyrexia (General disorders) | 6 (13) | 22 (29) | 9 (12) | 0 (0) | 2 (2) | 2 (4) | 0 | 0 | 0
Fatigue (General disorders) | 13 (25) | 5 (12) | 11 (26) | 4 (5) | 1 (2) | 2 (2) | 0 | 0 | 1
Chills (General disorders) | 11 (26) | 9 (27) | 5 (11) | 0 (0) | 2 (4) | 0 (0) | 0 | 0 | 0
Asthenia (General disorders) | 9 (11) | 6 (9) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 17 (21) | 23 (30) | 22 (49) | 2 (2) | 1 (1) | 4 (4) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 17 (37) | 13 (19) | 20 (34) | 3 (6) | 1 (1) | 3 (3) | 0 | 0 | 1
Influenza (Infections and infestations) | 9 (12) | 10 (17) | 17 (20) | 2 (2) | 0 (0) | 2 (2) | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 9 (10) | 5 (9) | 10 (11) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 9 (19) | 6 (12) | 8 (18) | 1 (1) | 2 (7) | 1 (4) | 0 | 0 | 0
Headache (Nervous system disorders) | 46 (145) | 37 (129) | 46 (135) | 3 (20) | 2 (2) | 5 (14) | 1 | 0 | 2
Paresthesia (Nervous system disorders) | 7 (16) | 8 (17) | 16 (27) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 12 (21) | 11 (17) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 6 (7) | 10 (12) | 6 (9) | 2 (2) | 1 (1) | 0 (0) | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 4 (5) | 4 (5) | 9 (9) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Depression (Psychiatric disorders) | 14 (17) | 9 (10) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 10 (10) | 7 (21) | 14 (20) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 14 (15) | 11 (12) | 5 (6) | 3 (3) | 3 (3) | 3 (3) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 10 (11) | 9 (10) | 3 (3) | 3 (3) | 1 (1) | 4 (4) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (13) | 11 (14) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 13 (15) | 6 (7) | 1 (1) | 0 (0) | 2 (2) | 3 (5) | 0 | 0 | 0
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 2 (4) | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (6) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anti-thyroid antibody positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to publish any results communication in connection with the study. The PI shall submit any communications including study results to the sponsor for review 30 working days prior to communication submission. The sponsor can request the PI to modify or delete any sponsor's proprietary information. If the PI refuses the modification, the submission shall be postponed for 60 days from PI refusal, to provide the sponsor the opportunity to file a patent or seek legal remedies.